CLINICAL TRIAL: NCT05986370
Title: The METRIC Study Protocol: an Explanatory Randomized Controlled Trial Investigating the Neurophysiological Mechanisms Underlying the Therapeutic Effects of Spinal Manipulative Therapy for Chronic Primary Low Back Pain
Brief Title: The METRIC Study Protocol
Acronym: METRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Mathieu Piché, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: METRIC
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low-back Pain
Keywords: chronic primary low back pain; spinal manipulative therapy; nociplastic pain; central sensitization; C-fibers; brain; electroencephalography
MeSH Terms: conditions — Nociplastic Pain | interventions — Manipulation, Spinal; Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lumbar spinal manipulative therapy (Experimental): Participants will receive spinal manipulative therapy (SMT) exclusively at dysfunctional lumbar segments. Participants will receive 36 SMT sessions over 12 weeks, 3 times per week, each session lasting ≈15 min. Spinal manipulation will be performed using the diversified technique. For each treatment, the SMT provider will perform two spinal manipulations, one on each side of the most painful lumbar vertebra. During spinal manipulations, participants will lay on their side and they will be instructed to inhale and exhale fully before each thrust.
  Interventions: Procedure: lumbar spinal manipulative therapy
- full spine spinal manipulative therapy (Experimental): Participants will receive spinal manipulative therapy (SMT) at dysfunctional spinal segments in the lumbar AND other spine regions. Participants will receive 36 spinal manipulative therapy (SMT) sessions over 12 weeks, 3 times per week, each session lasting ≈15 min. Spinal manipulation will be performed using the diversified technique. For each treatment, the SMT provider will perform a minimum of two spinal manipulations, one on each side of the most painful lumbar vertebra. Spinal manipulation will also be delivered at other dysfunctional spinal segments, based on clinical examination. During spinal manipulations, participants will lay prone, supine or on their side and they will be instructed to inhale and exhale fully before each thrust.
  Interventions: Procedure: full spine spinal manipulative therapy
- sham spinal manipulative therapy (Sham Comparator): Participants will receive 36 sham SMT sessions (3x/week for 12 weeks, each session ≈15 min). This will target dysfunctional segments in the lumbar and other spine regions. Three maneuvers will be used:
  * Ventral decubitus: 1 to 5 light and brief manual contacts (≈ 20 N and 5 s) will be applied and quickly released over the spinous process of dysfunctional vertebrae identified during clinical examination.
  * Dorsal decubitus: sections of the treatment table will be slightly raised or lowered (≈ 5 cm) and their lower limbs' position changed once or twice e.g., knees bent, hips internally or externally rotated. Each position maintained during ≈ 30 s.
  * Lateral decubitus: 1 to 5 impulses at the lowest setting of the Activator V instrument (Activator Methods Int. Ltd., Phoenix, Arizona, USA) will be applied on their gluteus and quadratus lumborum muscles. The position of the instrument will change after each impulse.
  Interventions: Procedure: sham spinal manipulative therapy
- no intervention (No Intervention): This fourth arm will comprise healthy volunteers (age/sex-matched to the participants in the test intervention - lumbar group) who will not receive any intervention. The main purpose of this fourth group is to provide reference values to interpret some results obtained in participants with chronic primary low back pain.

INTERVENTIONS:
Procedure: lumbar spinal manipulative therapy — Spinal manipulative therapy involves the application of spinal manipulation over several sessions. Spinal manipulation is defined as a high-velocity, low-amplitude thrust performed by a clinician to move a segment of the spine in a specific direction. This type of intervention often generates cavitation sounds (audible pops).
  Other Names: spinal manipulation; chiropractic adjustment; grade 5 spinal mobilization
  Arms: lumbar spinal manipulative therapy
Procedure: sham spinal manipulative therapy — Sham spinal manipulative therapy (sham SMT), was designed to be structurally equivalent to SMT, i.e., to attend to the same body regions with the same amount of contact as well as to have the same number, frequency and length of sessions. SMT and sham SMT will be provided by the same treatment provider and will appear to be similarly tailored to the participants' condition. Sham SMT does not share the component of interest of SMT, i.e., the activation of deep high-threshold mechanoreceptors via high-velocity, low-amplitude thrusts applied to the spine. Yet, it shares all the other components not of interest in this study that may contribute to the placebo response, such as therapeutic alliance, contextual factors, physical touch, and expectations. Furthermore, deception will be used to balance expectations and enhance blinding.
  Other Names: control intervention; sham control; sham treatment; placebo
  Arms: sham spinal manipulative therapy
Procedure: full spine spinal manipulative therapy — Spinal manipulative therapy involves the application of spinal manipulation over several sessions. Spinal manipulation is defined as a high-velocity, low-amplitude thrust performed by a clinician to move a segment of the spine in a specific direction. This type of intervention often generates cavitation sounds (audible pops).
  Other Names: spinal manipulation; chiropractic adjustment; grade 5 spinal mobilization
  Arms: full spine spinal manipulative therapy

SUMMARY:
The goal of this clinical trial is to test the effects of spinal manipulative therapy in individuals with chronic primary low back pain and determine the neurophysiological mechanisms underlying pain relief. The main questions it aims to answer are: • Is pain relief produced by spinal manipulative therapy in patients with chronic primary low back pain caused by a reduction of C-fiber-related nociceptive processing? • Are these effects greater when spinal manipulative therapy is applied to the whole spine where it is clinically indicated compared with lumbar spine only? • Are these effects greater after 36 treatments over 3 months compared with 12 treatments over 1 month. Participants will receive spinal manipulative therapy (all clinically indicated spine segments or back only) or a control intervention. A group of healthy volunteers will be recruited to assess secondary outcome measures over the same time period, as reference data for comparisons. Researchers will compare the two groups receiving spinal manipulative therapy to the group receiving the control intervention to see if clinical pain relief and the reduction of temporal summation of second pain (produced experimentally) is significantly greater with spinal manipulative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Duration of current low back pain (LBP) episode ≥ 6 months;
* Average LBP intensity during the last 7 days ≥ 3/10;
* (For healthy volunteers only) To be of the same sex and age (± 1 year) as a participant with low back pain.

Exclusion Criteria:

* Diagnosis of back conditions other than chronic primary LBP e.g., failed back surgery syndrome, spondylosis, spondylolisthesis, spinal stenosis, herniated disc, infection, etc.;
* Presence of pain in another body location that is more severe than the pain in the lower back;
* Presence of a neurological deficit i.e., sensation loss, muscle weakness, decreased deep tendon reflexes;
* Presence of contraindications to spinal manipulative therapy e.g., recent fracture, history of spinal surgery, cauda equina syndrome, inflammatory arthritis, taking anticoagulant medication, active cancer, moderate to severe osteoporosis, abdominal aortic aneurysm;
* Underwent surgery in the last 3 months;
* Pregnancy, ≤ 3 months post-partum or planning to get pregnant in the next 12 months;
* History of spinal manipulative therapy in the past 12 months;
* Scoliosis ≥ 20°;
* BMI ≥ 40;
* Insufficient language skills in French to complete the questionnaires;
* Open or pending litigation for LBP or seeking/receiving disability compensation;
* Diagnosis of an illness affecting the sensorimotor functions e.g., diabetes, multiple sclerosis, amyotrophic lateral sclerosis;
* Diagnosis of mental health disorders (with the exception of anxiety and depression);
* Current drug or alcohol dependence;
* Skin of type I on the Fitzpatrick scale;
* (For healthy volunteers only) Regular use of pain medication or usage in the 48 h prior to data collection;
* (For healthy volunteers only) History of chronic pain;
* (For healthy volunteers only) Acute pain on the days of data collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-09-29 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
low back pain intensity | baseline, 1- , 2-, 3-, 4-, 5-, 6-, 7-, 8-, 9-, 10-, 11-, 12-, 26-, 39-, 52- and 64-weeks post-randomization.
  In accordance with recommendations for chronic pain trials, participants will be instructed to rate the intensity of their LBP using a numerical rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain imaginable). As in the brief pain inventory (BPI), they will be instructed to rate their pain: 1) right now; 2) on average over the last 7 days; 3) at its worst over the last 7 days; 4) at its best over the last 7 days.
temporal summation of second pain | baseline, 4- and 12-weeks post-randomization.
  Participants will receive a total of 160 painful laser stimuli, 80 single-pulse stimuli and 80 pulse trains (3 pulses delivered at 0.67 Hz). After each stimulus, participants will be prompted to rate second pain with the display of a numerical pain rating scale. The pain ratings of single pulses will be subtracted from the pain ratings of pulse trains to estimate the intensity of the temporal summation of second pain.

SECONDARY OUTCOMES:
low back pain frequency and duration | baseline, 1- , 2-, 3-, 4-, 5-, 6-, 7-, 8-, 9-, 10-, 11-, 12-, 26-, 39-, 52- and 64-weeks post-randomization.
  A modified version of the pain frequency-severity-duration scale will be used. Participants will be instructed to answer these 3 questions:
  * Is the pain recurrent (it comes in episodes) or continuous (it is always present)?
  * How many days in the past week have you had low back pain? (0, 1, 2, 3, 4, 5, 6, 7 days; a higher score means a worse outcome)
  * On average, how many hours per day does the pain last? (0; 1-4; 5-8; 9-12; 13-16; 17-20; 21-24 hours; a higher score means a worse outcome)
Pressure pain thresholds (PPTs) | baseline, 4- and 12-weeks post-randomization.
  PPT will be measured using a handheld digital algometer (Wagner Pain TestTM FPX, Greenwich, Connecticut, USA) and a standardized protocol. The algometer will be applied perpendicularly to the skin of the first test location and the pressure increased at approximately 50 kPa/s until pain is reported by the participant. This procedure will be repeated three times at the same test location. The PPT will be the average of the values obtained during these 3 trials. The same procedures will be repeated at the two other test locations. PPT will be tested on three different body locations: 1) Over the spinous process of the most painful vertebra between L1 and S1; 2) On the right lower limb in the dermatome corresponding to the level of the most painful vertebra; 3) in the center of the right thenar eminence.
C-fiber-related brain responses | baseline, 4- and 12-weeks post-randomization.
  Electroencephalography (EEG) will be recorded using a 64-channel BrainVision system with active Ag-AgCl electrodes mounted on an actiCAP, according to the International 10-20 system (Brain Products, Gilching, Germany). Electrodes will be nose-referenced, and the ground will be set at FPz. Signals will be sampled at 500 Hz. Eye movements and blinks will be recorded using electrooculography (EOG). Electrode impedance will be kept below 20 kΩ. Closed eyes resting state EEG will be recorded for 5 min prior to laser stimuli for exploratory EEG analyses. EEG activity will be recorded continuously. The outcome of interest from laser-evoked-brain activity is the response evoked by C-fiber activation. Laser-evoked potentials (LEP) and event-related spectral perturbations (ERSP) will be analyzed using validated methods.
Oswestry Disability Index (ODI) | baseline, 4-, 12-, 26-, 39-, 52- and 64-weeks post-randomization.
  Self-reported low back pain related disability will be evaluated using the French-Canadian version of the ODI (0-100%; a higher score means a worse outcome).
Back performance scale (BPS) | baseline, 4- and 12-weeks post-randomization.
  The BPS will be used as a performance based outcome of physical function. It includes five daily activities such as putting socks on or picking something on the floor (see PMID: 12444880 for more details). Each activity is rated from 0 to 3, and the five scores are added up (min = 0, max = 15; a higher score means a worse outcome).
Five times sit-to-stand test | baseline, 4- and 12-weeks post-randomization.
  The five times sit-to-stand test will be used as performance based outcome of physical function. Participant sitting on a supported chair will be instructed to stand and sit again as fast as possible, five times in a row. Time will be measured in seconds. The test will be performed twice and the average time for the two trials will be recorded (a higher score means a worse outcome).
Depression | baseline, 4- and 12-weeks post-randomization.
  Depression levels will be measured using the French-Canadian version of the Beck Depression Inventory (BDI; min = 0, max = 63; a higher score means a worse outcome).
Anxiety | baseline, 4- and 12-weeks post-randomization.
  Anxiety levels will be measured using the French-Canadian version of the State-Trait Anxiety Inventory, version Y (STAI-Y; min = 20, max = 80; a higher score means a worse outcome).
Pain catastrophizing | baseline, 4- and 12-weeks post-randomization.
  The main elements contributing to the pain experience according to the fear avoidance model of pain will be measured. Pain catastrophizing will be measured with the French-Canadian version of the pain catastrophizing scale (PCS; min = 0, max = 52; a higher score means a worse outcome).
Kinesiophobia | baseline, 4- and 12-weeks post-randomization.
  The main elements contributing to the pain experience according to the fear avoidance model of pain will be measured. Pain-related fear will be measured with a French adaptation of the Tampa scale for kinesiophobia (TSK; min = 17, max = 68; a higher score means a worse outcome).
Pain vigilance | baseline, 4- and 12-weeks post-randomization.
  The main elements contributing to the pain experience according to the fear avoidance model of pain will be measured. Hypervigilance will be measured with a French adaptation of the pain vigilance and awareness questionnaire (PVAQ; min = 0, max = 80; a higher score means a worse outcome).
Patient's global impression of change | After the last treatment session (12-weeks post-randomization)
  Participants will be instructed to give their global impression of change on a scale from -100 to 100 (-100 = very much worse, 0 = no change, 100 = very much improved).
Expectations of pain relief | baseline and 4-weeks post-randomization.
  Participants will be instructed to rate their expectations of pain relief after the treatment on a scale from 0 to 100, 0 being "no relief" and 100 being "complete relief".
Contextual factors (healing encounters and attitudes lists (HEAL)) | baseline, 4- and 12-weeks post-randomization.
  Contextual factors will be measured using a French adaptation of the healing encounters and attitudes lists (HEAL).

OTHER OUTCOMES:
Adverse events (AE) | 1- , 2-, 3-, 4-, 5-, 6-, 7-, 8-, 9-, 10-, 11-, 12-, 13-weeks post-randomization.
  Participants will be informed of the risk of AE and the importance to communicate any unpleasant or abnormal sensation occurring in the hours or days following a treatment. Mild AE are defined as transient reactions (≤ 48 h) that do not require further treatment. Moderate AE are defined as reactions lasting more than 48 h, limiting function or daily activity and possibly requiring additional care. Severe AE are defined as reactions requiring hospital admission, life threatening, or causing long-lasting disability.
Blinding | After the last treatment session (12-weeks post-randomization)
  Blinding will be assessed by asking these questions: 1) Do you think that you received a real chiropractic treatment for low back pain? (yes / no) 2) How certain are you on a scale of 0 to 10, where 0 indicates certainty of not having received a chiropractic treatment, 5 indicates absolute uncertainty, and 10 absolute certainty of having received a chiropractic treatment
Number of other treatments for low back pain | 1- , 2-, 3-, 4-, 5-, 6-, 7-, 8-, 9-, 10-, 11-, 12-weeks post-randomization.
  Participants will be informed about the possibility to seek care for their low back pain outside the study at any point, if necessary. Based on recent Canadian practice guidelines for chronic LBP, exercise and oral nonsteroidal anti-inflammatory drugs (NSAIDs) will be recommended as first alternatives to interventions provided in the study. However, participants may receive other treatments. The number of concomitant treatments will be measured once a week by asking these questions:
  * In the past 7 days, have you used or received any other treatment for low back pain than the one provided in this study? (yes / no)
  * If so, please specify the number of treatments you received (for example: the number of pills taken, the number of therapy sessions, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Piché, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
After publication of the results, the data that support the findings of this study will be available from the corresponding author, MP, upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon publication of the results (expected in January 2026). They will be available for the next 5 years.

REFERENCES:
- [Background] Buchbinder R, Underwood M, Hartvigsen J, Maher CG. The Lancet Series call to action to reduce low value care for low back pain: an update. Pain. 2020 Sep;161 Suppl 1(1):S57-S64. doi: 10.1097/j.pain.0000000000001869. No abstract available. PMID 33090740
- [Background] Cormier S, Lavigne GL, Choiniere M, Rainville P. Expectations predict chronic pain treatment outcomes. Pain. 2016 Feb;157(2):329-338. doi: 10.1097/j.pain.0000000000000379. PMID 26447703
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Chronic primary musculoskeletal pain: a new concept of nonstructural regional pain. Pain Rep. 2022 Aug 9;7(5):e1024. doi: 10.1097/PR9.0000000000001024. eCollection 2022 Sep-Oct. PMID 35975135
- [Background] Funabashi M, Gorrell LM, Pohlman KA, Bergna A, Heneghan NR. Definition and classification for adverse events following spinal and peripheral joint manipulation and mobilization: A scoping review. PLoS One. 2022 Jul 15;17(7):e0270671. doi: 10.1371/journal.pone.0270671. eCollection 2022. PMID 35839253
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Gevers-Montoro C, Provencher B, Descarreaux M, Ortega de Mues A, Piche M. Neurophysiological mechanisms of chiropractic spinal manipulation for spine pain. Eur J Pain. 2021 Aug;25(7):1429-1448. doi: 10.1002/ejp.1773. Epub 2021 Apr 15. PMID 33786932
- [Background] Gevers-Montoro C, Provencher B, Northon S, Stedile-Lovatel JP, Ortega de Mues A, Piche M. Chiropractic Spinal Manipulation Prevents Secondary Hyperalgesia Induced by Topical Capsaicin in Healthy Individuals. Front Pain Res (Lausanne). 2021 Jul 20;2:702429. doi: 10.3389/fpain.2021.702429. eCollection 2021. PMID 35295504
- [Background] Graven-Nielsen T. Mechanisms and manifestations in musculoskeletal pain: from experimental to clinical pain settings. Pain. 2022 Nov 1;163(Suppl 1):S29-S45. doi: 10.1097/j.pain.0000000000002690. Epub 2022 May 15. No abstract available. PMID 35984370
- [Background] Greco CM, Yu L, Johnston KL, Dodds NE, Morone NE, Glick RM, Schneider MJ, Klem ML, McFarland CE, Lawrence S, Colditz J, Maihoefer CC, Jonas WB, Ryan ND, Pilkonis PA. Measuring nonspecific factors in treatment: item banks that assess the healthcare experience and attitudes from the patient's perspective. Qual Life Res. 2016 Jul;25(7):1625-34. doi: 10.1007/s11136-015-1178-1. Epub 2015 Nov 12. PMID 26563249
- [Background] Haas M, Vavrek D, Peterson D, Polissar N, Neradilek MB. Dose-response and efficacy of spinal manipulation for care of chronic low back pain: a randomized controlled trial. Spine J. 2014 Jul 1;14(7):1106-16. doi: 10.1016/j.spinee.2013.07.468. Epub 2013 Oct 16. PMID 24139233
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hohenschurz-Schmidt D, Vase L, Scott W, Annoni M, Ajayi OK, Barth J, Bennell K, Berna C, Bialosky J, Braithwaite F, Finnerup NB, Williams ACC, Carlino E, Cerritelli F, Chaibi A, Cherkin D, Colloca L, Cote P, Darnall BD, Evans R, Fabre L, Faria V, French S, Gerger H, Hauser W, Hinman RS, Ho D, Janssens T, Jensen K, Johnston C, Juhl Lunde S, Keefe F, Kerns RD, Koechlin H, Kongsted A, Michener LA, Moerman DE, Musial F, Newell D, Nicholas M, Palermo TM, Palermo S, Peerdeman KJ, Pogatzki-Zahn EM, Puhl AA, Roberts L, Rossettini G, Tomczak Matthiesen S, Underwood M, Vaucher P, Vollert J, Wartolowska K, Weimer K, Werner CP, Rice ASC, Draper-Rodi J. Recommendations for the development, implementation, and reporting of control interventions in efficacy and mechanistic trials of physical, psychological, and self-management therapies: the CoPPS Statement. BMJ. 2023 May 25;381:e072108. doi: 10.1136/bmj-2022-072108. No abstract available. PMID 37230508
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] Korownyk CS, Montgomery L, Young J, Moore S, Singer AG, MacDougall P, Darling S, Ellis K, Myers J, Rochford C, Taillefer MC, Allan GM, Perry D, Moe SS, Ton J, Kolber MR, Kirkwood J, Thomas B, Garrison S, McCormack JP, Falk J, Dugre N, Sept L, Turgeon RD, Paige A, Potter J, Nickonchuk T, Train AD, Weresch J, Chan K, Lindblad AJ. PEER simplified chronic pain guideline: Management of chronic low back, osteoarthritic, and neuropathic pain in primary care. Can Fam Physician. 2022 Mar;68(3):179-190. doi: 10.46747/cfp.6803179. PMID 35292455
- [Background] Kosek E, Clauw D, Nijs J, Baron R, Gilron I, Harris RE, Mico JA, Rice ASC, Sterling M. Chronic nociplastic pain affecting the musculoskeletal system: clinical criteria and grading system. Pain. 2021 Nov 1;162(11):2629-2634. doi: 10.1097/j.pain.0000000000002324. No abstract available. PMID 33974577
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] McPhee ME, Vaegter HB, Graven-Nielsen T. Alterations in pronociceptive and antinociceptive mechanisms in patients with low back pain: a systematic review with meta-analysis. Pain. 2020 Mar;161(3):464-475. doi: 10.1097/j.pain.0000000000001737. PMID 32049888
- [Background] Mucke M, Cuhls H, Radbruch L, Baron R, Maier C, Tolle T, Treede RD, Rolke R. Quantitative sensory testing (QST). English version. Schmerz. 2021 Nov;35(Suppl 3):153-160. doi: 10.1007/s00482-015-0093-2. PMID 26826097
- [Background] Nicholas M, Vlaeyen JWS, Rief W, Barke A, Aziz Q, Benoliel R, Cohen M, Evers S, Giamberardino MA, Goebel A, Korwisi B, Perrot S, Svensson P, Wang SJ, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic primary pain. Pain. 2019 Jan;160(1):28-37. doi: 10.1097/j.pain.0000000000001390. PMID 30586068
- [Background] Nijs J, Apeldoorn A, Hallegraeff H, Clark J, Smeets R, Malfliet A, Girbes EL, De Kooning M, Ickmans K. Low back pain: guidelines for the clinical classification of predominant neuropathic, nociceptive, or central sensitization pain. Pain Physician. 2015 May-Jun;18(3):E333-46. PMID 26000680
- [Background] Nim CG, Kawchuk GN, Schiottz-Christensen B, O'Neill S. The effect on clinical outcomes when targeting spinal manipulation at stiffness or pain sensitivity: a randomized trial. Sci Rep. 2020 Sep 3;10(1):14615. doi: 10.1038/s41598-020-71557-y. PMID 32884045
- [Background] Ozudogru A, Canli M, Ceylan I, Kuzu S, Alkan H, Karacay BC. Five Times Sit-to-Stand Test in people with non-specific chronic low back pain-a cross-sectional test-retest reliability study. Ir J Med Sci. 2023 Aug;192(4):1903-1908. doi: 10.1007/s11845-022-03223-3. Epub 2022 Nov 15. PMID 36376556
- [Background] Plaghki L, Mouraux A. How do we selectively activate skin nociceptors with a high power infrared laser? Physiology and biophysics of laser stimulation. Neurophysiol Clin. 2003 Dec;33(6):269-77. doi: 10.1016/j.neucli.2003.10.003. PMID 14678841
- [Background] Plaghki L, Mouraux A. EEG and laser stimulation as tools for pain research. Curr Opin Investig Drugs. 2005 Jan;6(1):58-64. PMID 15675604
- [Background] Provencher B, Northon S, Gevers Montoro C, O'Shaughnessy J, Piche M. Effects of chiropractic spinal manipulation on laser-evoked pain and brain activity. J Physiol Sci. 2021 Jun 24;71(1):20. doi: 10.1186/s12576-021-00804-2. PMID 34167458
- [Background] Provencher B, Northon S, Piche M. Segmental Chiropractic Spinal Manipulation Does not Reduce Pain Amplification and the Associated Pain-Related Brain Activity in a Capsaicin-Heat Pain Model. Front Pain Res (Lausanne). 2021 Nov 1;2:733727. doi: 10.3389/fpain.2021.733727. eCollection 2021. PMID 35295444
- [Background] Puhl AA, Reinhart CJ, Doan JB, Vernon H. The quality of placebos used in randomized, controlled trials of lumbar and pelvic joint thrust manipulation-a systematic review. Spine J. 2017 Mar;17(3):445-456. doi: 10.1016/j.spinee.2016.11.003. Epub 2016 Nov 22. PMID 27888138
- [Background] Schaffler K, Nicolas LB, Borta A, Brand T, Reitmeir P, Roebling R, Scholpp J. Investigation of the predictive validity of laser-EPs in normal, UVB-inflamed and capsaicin-irritated skin with four analgesic compounds in healthy volunteers. Br J Clin Pharmacol. 2017 Jul;83(7):1424-1435. doi: 10.1111/bcp.13247. Epub 2017 Feb 27. PMID 28139023
- [Background] Shraim MA, Masse-Alarie H, Hall LM, Hodges PW. Systematic Review and Synthesis of Mechanism-based Classification Systems for Pain Experienced in the Musculoskeletal System. Clin J Pain. 2020 Oct;36(10):793-812. doi: 10.1097/AJP.0000000000000860. PMID 32852923
- [Background] Starkweather AR, Heineman A, Storey S, Rubia G, Lyon DE, Greenspan J, Dorsey SG. Methods to measure peripheral and central sensitization using quantitative sensory testing: A focus on individuals with low back pain. Appl Nurs Res. 2016 Feb;29:237-41. doi: 10.1016/j.apnr.2015.03.013. Epub 2015 Apr 8. PMID 26856520
- [Background] Stevans JM, Delitto A, Khoja SS, Patterson CG, Smith CN, Schneider MJ, Freburger JK, Greco CM, Freel JA, Sowa GA, Wasan AD, Brennan GP, Hunter SJ, Minick KI, Wegener ST, Ephraim PL, Friedman M, Beneciuk JM, George SZ, Saper RB. Risk Factors Associated With Transition From Acute to Chronic Low Back Pain in US Patients Seeking Primary Care. JAMA Netw Open. 2021 Feb 1;4(2):e2037371. doi: 10.1001/jamanetworkopen.2020.37371. PMID 33591367
- [Background] Strand LI, Moe-Nilssen R, Ljunggren AE. Back Performance Scale for the assessment of mobility-related activities in people with back pain. Phys Ther. 2002 Dec;82(12):1213-23. PMID 12444880
- [Background] Verdugo RJ, Matamala JM, Inui K, Kakigi R, Valls-Sole J, Hansson P, Nilsen KB, Lombardi R, Lauria G, Petropoulos IN, Malik RA, Treede RD, Baumgartner U, Jara PA, Campero M. Review of techniques useful for the assessment of sensory small fiber neuropathies: Report from an IFCN expert group. Clin Neurophysiol. 2022 Apr;136:13-38. doi: 10.1016/j.clinph.2022.01.002. Epub 2022 Jan 19. PMID 35131635
- [Background] Vlaeyen JWS, Crombez G, Linton SJ. The fear-avoidance model of pain. Pain. 2016 Aug;157(8):1588-1589. doi: 10.1097/j.pain.0000000000000574. No abstract available. PMID 27428892
- [Background] Wheeler CHB, Williams ACC, Morley SJ. Meta-analysis of the psychometric properties of the Pain Catastrophizing Scale and associations with participant characteristics. Pain. 2019 Sep;160(9):1946-1953. doi: 10.1097/j.pain.0000000000001494. PMID 30694929
- [Background] Wang YP, Gorenstein C. Psychometric properties of the Beck Depression Inventory-II: a comprehensive review. Braz J Psychiatry. 2013 Oct-Dec;35(4):416-31. doi: 10.1590/1516-4446-2012-1048. Epub 2013 Dec 23. PMID 24402217
- [Background] Denis I, Fortin L. Development of a French-Canadian version of the Oswestry Disability Index: cross-cultural adaptation and validation. Spine (Phila Pa 1976). 2012 Apr 1;37(7):E439-44. doi: 10.1097/BRS.0b013e318233eaf9. PMID 22037523
- [Background] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT05986370/SAP_000.pdf